CLINICAL TRIAL: NCT04178109
Title: EVALUATION OF ORAL USE OF DEXKETOPROFEN/TRAMADOL IN ACUTE POSTOPERATIVE PAIN IN PATIENTS UNDERGOING TOTAL HIP REPLACEMENT WITH A MINIMALLY INVASIVE ANTERIOR APPROACH (AMIS).
Brief Title: Oral Use of Dexketoprofen/Tramadol for Acute Postoperative Pain in Total Hip Replacement With a Direct Anterior Approach.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KAT General Hospital (Other)
Responsible Party: Principal Investigator, Elena Nikolakopoulou, MD, KAT General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17200
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Pain; Pain, Acute
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — dexketoprofen trometamol; Tramadol; Acetaminophen; Ropivacaine; Levobupivacaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A was under spinal anesthesia with a 25G cutting edge needle with levobupivacaine 10-15mg and fentanyl 10μg.
  Periarticular injection was done by the surgeon with a dilition of 100ml N/S 0,9% with 300mg ropivacaine and 0,5mg epinephrine.
  Group A was given the oral combination dexketoprofen/tramadole (25mg/75mg) 2h after surgery every 8h for 72h.
  Interventions: Drug: Dexketoprofen/tramadol (27mg/75mg); Drug: Ropivacaine Hydrochloride 7.5 MG/ML; Drug: Levobupivacaine Hydrochloride
- Group B (Placebo Comparator): Group B was under spinal anesthesia with a 25G cutting edge needle with levobupivacaine 10-15mg and fentanyl 10μg.
  Periarticular injection was done by the surgeon with a dilition of 100ml N/S 0,9% with 300mg ropivacaine and 0,5mg epinephrine.
  Group B received postoperative analgesia with intravenous tramadole 75mg and paracetamol 1g every 8h with the first dose beginning 2h after the end of the surgery. For 72h
  Interventions: Drug: Tramadol hydrochloride; Drug: Paracetamol; Drug: Ropivacaine Hydrochloride 7.5 MG/ML; Drug: Levobupivacaine Hydrochloride

INTERVENTIONS:
Drug: Dexketoprofen/tramadol (27mg/75mg) — Postoperatively patients in Group A received the oral combination dexketoprofen/tramadol for the treatment of acute postoperative pain the first 72h
  Arms: Group A
Drug: Tramadol hydrochloride — Patients in group B received IV tramadol 75mg every 8h
  Arms: Group B
Drug: Paracetamol — Patients in group B received IV paracetamol 1g every 8h
  Arms: Group B
Drug: Ropivacaine Hydrochloride 7.5 MG/ML — 300mg ropivacaine as periarticular injection in a dilution of 100ml n/s 0,9% was done by the orthopedic surgeon in all patients
Drug: Levobupivacaine Hydrochloride — 10-15mg levobupivacaine was done subarachnoidal for spinal anesthesia

SUMMARY:
Pain is a global public health issue and represents the most common reason for both physician consultation and hospital admissions . When unrelieved or poorly controlled, it is associated with medical complications, poor patient satisfaction and increased risk of developing chronic pain. Dexketoprofen is a new NSAID treating acute postoperative pain and when it combined with tramadol may have a better effect. The purpose of this study is to evaluate the analgesic effect of the oral use of the combination of dexketoprofen/tramadole on the reduction of postoperative pain after total hip arthroplasty with minimal invasive anterior approach (AMIS).

ELIGIBILITY:
Inclusion Criteria:

* unilateral total hip arthroplasty with a direct anterior minimal invasive technique
* ASA score I or II
* signed written informed consent form
* 3 days hospitalization
* 45-80 years old
* primary Total hip arthroplasty

Exclusion Criteria:

* allergy to any given drugs
* contraindications for spinal anesthesia
* active bleeding
* renal failure ( gfr< 90ml/h)
* hepatic failure ( abnormal sgot,sgpt,γgt)
* heart failure
* history of gastrointestinal bleeding

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Pain score in 8hours | 8 hours
  Pain score with the visualised analogue scale in 8hours
Pain score in 24hours | 24 hours
  Pain score with the visualised analogue scale in 24 hours
Pain score in 48 hours | 48 hours
  Pain score with the visualised analogue scale in 48 hours
Pain score in 72 hours | 72 hours
  Pain score with the visualised analogue scale in 72 hours
Total analgesic consumption | 24 houra
  Total analgesic consumption as rescue analgesia the first 24 hours

SECONDARY OUTCOMES:
Side effects | 72 hours
  All the side effects of the drug the first 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Elena Nikolakopoulou, Athens, Kifissia, Greece

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Macheras GA, Tzefronis D, Argyrou C, Nikolakopoulou E, Galvez Miravete A, Karachalios TS. Pain management after total hip arthroplasty: comparative study of analgesic efficacy and tolerability between oral tramadol/dexketoprofen and injectable paracetamol + tramadol. Hip Int. 2024 May;34(3):304-310. doi: 10.1177/11207000231219797. Epub 2024 Jan 10. PMID 38204364